CLINICAL TRIAL: NCT04658641
Title: Characterization of Complex Pulse Shapes in Deep Brain Stimulation for Movement Disorders Using EEG and Local Field Potential Recordings
Acronym: CHANNEL DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Myles Mc Laughlin, Prof. Dr. Myles Mc Laughlin, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: S62373
Record Dates: First submitted 2020-11-24; First posted 2020-12-08 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Parkinson Disease; Essential Tremor
MeSH Terms: conditions — Parkinson Disease; Essential Tremor

STUDY DESIGN:
Intervention Model Description: Randomized, crossover, blinded design
Who Masked: Participant
Masking Description: Blinded design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard clinical pulse shape (Active Comparator): Standard clinical pulse shape as used in clinical practice (cathodic stimulation).
  Interventions: Device: Boston Scientific: Study tool computer
- Complex pulse shape (Experimental): Complex pulse shape (i.e. biphasic pulse shape anode first, biphasic pulse shape cathode first, hyperpolarizing pre-pulse or depolarizing pre-pulse).
  Interventions: Device: Boston Scientific: Study tool computer

INTERVENTIONS:
Device: Boston Scientific: Study tool computer — Compare clinical outcome measurements of complex pulse shapes to standard clinical pulse shape

SUMMARY:
Parkinson's disease and essential tremor are chronic movement disorders for which there is no cure. When medication is no longer effective, deep brain stimulation (DBS) is recommended. Standard DBS is a neuromodulation method that uses a simple monophasic pulse, delivered from an electrode to stimulate neurons in a target brain area. This monophasic pulse spreads out from the electrode creating a broad, electric field that stimulates a large neural population. This can often effectively reduce motor symptoms. However, many DBS patients experience side effects - caused by stimulation of non-target neurons - and suboptimal symptom control - caused by inadequate stimulation of the correct neural target. The ability to carefully manipulate the stimulating electric field to target specific neural subpopulations could solve these problems and improve patient outcomes. The use of complex pulse shapes, specifically biphasic pulses and asymmetric pre-pulses, can control the temporal properties of the stimulation field. Evidence suggests that temporal manipulations of the stimulation field can exploit biophysical differences in neurons to target specific subpopulations. Therefore, our aim is to evaluate the direct neurophysiological effects of complex pulse shapes in DBS movement disorder patients. This will be achieved using a two-stage investigation: stage one will study the neural response to different pulse shapes using electroencephalography (EEG) recordings. Stage two will study the neural responses to different pulse shapes using intra-operative local field potential (LFP) recordings. This study only relates only to the collection of EEG and LFP recordings in DBS patients. The protocol does not cover any surgical procedures, which already take place as part of the patient's normal clinical care.

DETAILED DESCRIPTION:
Parkinson's disease and essential tremor are chronic movement disorders for which there is no cure. When medication is no longer effective, deep brain stimulation (DBS) is recommended. Standard DBS is a neuromodulation method that uses a simple monophasic pulse, delivered from an electrode to stimulate neurons in a target brain area. This monophasic pulse spreads out from the electrode creating a broad, electric field that stimulates a large neural population. This can often effectively reduce motor symptoms. However, many DBS patients experience side effects - caused by stimulation of non-target neurons - and suboptimal symptom control - caused by inadequate stimulation of the correct neural target. The ability to carefully manipulate the stimulating electric field to target specific neural subpopulations could solve these problems and improve patient outcomes.

It has been shown that modifying the electrical waveform (e.g. pulse duration, pulse polarity, etc.) determine the spatial selectivity in functional electrical stimulation. Also, a recent clinical study examined for the first time the acute effects of anodic compared to cathodic neurostimulation in 10 PD patients. They found that thresholds for anodic stimulation were significantly higher than thresholds for cathodic stimulation, which is in agreement with previous research in animal studies and model calculations. However, they also reported a better clinical effect of anodic compared to cathodic stimulation. Furthermore, a modeling study from Anderson et al. (2018) found that fiber orientations can be selectively targeted depending on the stimulus waveform (i.e. cathodic or anodic). Another recent study examined the effect of an active symmetric biphasic pulse in 8 PD and 3 ET patients. They found that this pulse shapes produced significant clinical improvements compared to the standard clinical pulse shape.

Besides the symmetric biphasic pulse shape, the asymmetric pre-pulse shows great potential for the refinement of DBS therapy. If the pre-pulse is anodic, it has a hyperpolarizing effect and is therefore referred to as a hyperpolarizing pre-pulse. If it is cathodic, it has a depolarizing effect near the electrode and is therefore referred to as a depolarizing pre-pulse. Clinical studies focused on the use of asymmetric pulse shapes to improve the spatial selectivity by selectively exciting fibers in cochlear implant listeners13-16. Modeling studies indicate that a hyperpolarizing pre-pulse can actually decrease the threshold for axons and that the threshold is decreased more for axons close to the electrode than axons further away. This indicates that a hyperpolarizing pre-pulse may help focus the effects of stimulation to axons near the electrode, thus leading to an increase in the therapeutic window and potentially more efficient symptom control.

Evidence suggests that temporal manipulations (i.e. the use of complex pulse shapes, specifically biphasic pulses and asymmetric pre-pulses) of the stimulation field can exploit biophysical differences in neurons to target specific subpopulations. Ultimately, this may lead to an increase in the therapeutic window and/or more efficient symptom control. In this study, we aim to understand the neural mechanism underpinning the clinical effects observed by manipulating the pulse shapes, by comparing neurophysiological responses to the standard clinical pulse shapes to the responses to the complex pulse shapes. This will be achieved using two approaches. The first approach will study neural responses to different pulse shapes using electroencephalography (EEG) recordings. The second approach will study neural responses to different pulse shapes using intra-operative local field potential (LFP) recordings. This study and research protocol relates only to the collection of EEG and LFP recordings in DBS patients. The protocol does not cover any surgical procedures, which will already take place as part of the patient's normal clinical care.

ELIGIBILITY:
Inclusion Criteria for PD:

* Diagnosis of idiopathic Parkinson's disease where the diagnosis was made by a Movement Disorder Specialist according to the MDS criteria of 2015, with a Hoehn and Yahr scale (H&Y) of at least 2 (bilateral involvement).
* Onset of the symptoms more than five years ago.
* MDS-UPDRS-III score of ≥30 without medication or DBS.
* Electrodes are implanted in target area STN.

Inclusion Criteria for ET:

* Patient is diagnosed with essential tremor by a Movement Disorder Specialist.
* Diagnosis since more than 3 years.
* Patient has a disabling medical-refractory upper extremity tremor without medication or DBS.
* Patient has a postural or kinetic tremor severity score of at least 3 out of 4 in the extremity intended for treatment on the Fahn-Tolosa-Marin Clinical Rating Scale for Tremor without medication or DBS.
* Electrodes are implanted in target area VIM.

General Inclusion Criteria:

Post-op the implanted electrodes pass an integrity check, i.e. no open or shorted electrodes.

* Stable medications
* Lack of dementia or depression.
* Patient is willing and able to comply with all visits and study related procedures
* Patient understands the study requirements and the treatment procedures and provides written informed consent before any study-specific tests or procedures are performed.
* Patient can tolerate at least 12 hours OFF medication and per clinical judgement be able to perform all study related procedures

Exclusion Criteria:

* Any significant psychiatric problems, including unrelated clinically significant depression.
* Any current drug or alcohol abuse.
* Any history of recurrent or unprovoked seizures.
* Have any significant medical condition that is likely to interfere with study procedures or likely to confound evaluation of study endpoints, including any terminal illness with survival <12 months.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Peak height | During EEG/LFP recordings (approximately 1 hour per experiment)
  Extracted from EEG/LFP evoked potential responses
Peak timing | During EEG/LFP recordings (approximately 1 hour per experiment)
  Extracted from EEG/LFP evoked potential responses

CONTACTS AND LOCATIONS:
Overall Officials: Myles Mc Laughlin, Prof. Dr., Principal Investigator — KU Leuven; Bart Nuttin, Prof. Dr., Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Bogaert T, Peeters J, Boogers A, Vandenberghe W, De Vloo P, Nuttin B, Mc Laughlin M. Evoked Resonant Neural Activity Reveals an Electrophysiologic Sweet Spot for Directional Subthalamic Nucleus Deep Brain Stimulation in Parkinson's Disease. Neuromodulation. 2025 Oct 16:S1094-7159(25)01027-X. doi: 10.1016/j.neurom.2025.09.303. Online ahead of print. PMID 41099685
- [Derived] Peeters J, Boogers A, Van Bogaert T, Dembek TA, Gransier R, Wouters J, Vandenberghe W, De Vloo P, Nuttin B, Mc Laughlin M. Towards biomarker-based optimization of deep brain stimulation in Parkinson's disease patients. Front Neurosci. 2023 Jan 11;16:1091781. doi: 10.3389/fnins.2022.1091781. eCollection 2022. PMID 36711127
- [Derived] Peeters J, Boogers A, Van Bogaert T, Davidoff H, Gransier R, Wouters J, Nuttin B, Mc Laughlin M. Electrophysiologic Evidence That Directional Deep Brain Stimulation Activates Distinct Neural Circuits in Patients With Parkinson Disease. Neuromodulation. 2023 Feb;26(2):403-413. doi: 10.1016/j.neurom.2021.11.002. Epub 2021 Dec 18. PMID 35088733